CLINICAL TRIAL: NCT01865539
Title: Efficacy of Foot Orthotics in Veterans With Chronic Lower Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment/funding
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Collaborators: Foot Levelers, Inc. (Industry); Northeast College of Health Sciences (Other)
Responsible Party: Principal Investigator, Paul Dougherty, DC, Chiropractor, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIRB00558
Record Dates: First submitted 2013-05-20; First posted 2013-05-31 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Chronic lower back pain; Custom foot orthotics; Veterans

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custom Foot Orthotic (Active Comparator): Custom foot orthotic
  Interventions: Device: Custom Foot Orthotic
- Sham Orthotic (Sham Comparator): Will be a sham orthotic that will be the same as the actual orthotic without the custom support pads.
  Interventions: Device: Sham Orthotic

INTERVENTIONS:
Device: Custom Foot Orthotic — Custom foot orthotic with custom design pads
  Other Names: Foot Levelers Custom Foot Orthotic
  Arms: Custom Foot Orthotic
Device: Sham Orthotic — Leather insert without the custom design pads
  Arms: Sham Orthotic

SUMMARY:
A randomized sham controlled trial evaluating the efficacy of the use of custom foot orthotics in veterans suffering from chronic lower back pain. The current study hypothesizes that those veterans with chronic lower back pain who receive the custom foot orthotics will show greater improvements in pain and disability associated with the chronic lower back pain than those who receive the sham orthotic.

DETAILED DESCRIPTION:
Specific Aim 1: Utilizing a gold standard sham controlled randomized trial design, we will evaluate the change in pain, back related disability and quality of life in Veterans with chronic lower back pain who utilize either a custom foot orthotic or a sham orthotic.

As part of this aim the investigators will build on the teams strength of recruiting and enrolling Veteran's with chronic lower back pain into a randomized trial. The investigators will collect baseline pain and disability measures utilizing validated tools. Once the patients are enrolled, utilizing the "gold standard" placebo controlled design the investigators will randomize patients to receive either a custom foot orthotic or a sham orthotic. The Veterans will then be assessed at 5, 12 and 24-weeks post baseline to evaluate differences in pain and disability. Based on previous studies on the effectiveness of custom foot orthotics the investigators hypothesize that that Veteran's who receive the custom orthotic will experience less pain and disability as compared to those who receive the sham orthotics.

Specific Aim 2: To evaluate baseline characteristics of Veterans with chronic lower back pain predictive of responsiveness to custom foot orthotics including age, BMI, psychosocial characteristics and arch classification.

Focusing on the Veterans who receive the custom foot orthotic, the investigators next examine the important characteristics that may predict those Veterans who are most likely to benefit from wearing custom foot orthotics. Assessing potential confounders or facilitators of effectiveness of the custom foot orthotic will allow the investigators to best describe potential mechanisms of responsiveness. The investigators have chosen previously described confounders to responsiveness to treatment of chronic lower back pain, specifically age, body mass index and psychosocial characteristics. This methodology is particularly important in a sham controlled trial to assess if effectiveness or lack of thereof, is a factor of the intervention or from other confounding variables. The investigators have also chosen to evaluate the arch classification based on the measurement of the Veterans arch; again this allows for specific recommendations concerning use of this product. Based on previous studies on the effectiveness of custom foot orthotics in addition to previous studies evaluating chronic lower back pain the investigators hypothesize that those Veterans who are older, have a higher BMI and greater fear avoidance belief scores will show less responsiveness to the custom foot orthotics as compared to those younger Veterans who have a lower BMI and lower fear avoidance belief scores. In addition based on previous biomechanical literature, the investigators feel that those Veterans with a lower arch will show the greatest responsiveness to the custom foot orthotic.

ELIGIBILITY:
INCLUSION:

Ages 18-65 Lower back pain ≥ 3 months in duration Pain elicited upon deep palpation of the lumbar erector spinae musculature Primary complaint of CLBP from L1 to Sacroiliac joint inclusive. Ability/willingness to use orthotics in their shoes Numeric Pain Rating Scale (NRPS) of ≥ 3

* 30 mm on the Visual Analogue Scale (VAS)
* 20% for the Modified Oswestry Disability Index (mODI)

EXCLUSION:

spinal surgery, spinal injections or injections in their feet within the past 6 months Inability to use orthotics in shoes Custom foot orthotics within the past 12 months Currently undergoing Chiropractic, Physical Therapy or Acupuncture treatment for their chronic lower back pain.

evidence of cauda equina syndrome, spinal neoplasia or metastatic disease, destructive joint pathology such as rheumatoid arthritis bowel/bladder dysfunction (associated with the back pain) peripheral neuropathy or progressive lumbosacral radiculopathy, progressive myelopathy or neurogenic claudication.

open workers compensation or no fault case.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Dougherty, DC, Principal Investigator — Canandaigua VA Medical Center/ New York Chiropractic College
Locations (1):
- Rochester Outpatient Clinic (ROPC) of the Canandaigua VA Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahar T, Cohen MJ, Uval-Ne'eman V, Kandel L, Odebiyi DO, Lev I, Brezis M, Lahad A. Insoles for prevention and treatment of back pain: a systematic review within the framework of the Cochrane Collaboration Back Review Group. Spine (Phila Pa 1976). 2009 Apr 20;34(9):924-33. doi: 10.1097/BRS.0b013e31819f29be. PMID 19359999
- See also: New York Chiropractic College — http://www.nycc.edu
- See also: Foot Levelers Website — http://www.footlevelers.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Custom Foot Orthotic | Sham Orthotic
Started | 21 | 30
Completed | 21 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom Foot Orthotic | Sham Orthotic | Total
Number analyzed (Participants) | 21 | 30 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 30 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.1) | 55.1 (10.5) | 56.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 20 | 26 | 46
Region of Enrollment [Number; unit: participants]
  United States | 21 | 30 | 51

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: Visual Analog Scales (VAS): VAS is rated from 0 to 100mm with 0 being no pain at all and 100mm being the worst pain imaginable. The test has shown test-retest reliability, intra-examiner reliability and inter-examiner reliability.
Time Frame: 24 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Foot Orthotic | Sham Orthotic
Number analyzed (Participants) | 21 | 30
units on a scale | 57.7 (15.6) | 59.2 (14.9)

2. Secondary Outcome: Modified Oswestry Disability Index (mODI)
Description: The back pain specific, self-rating scale evaluates the degree of functional impairment that a patient is experiencing in a number of activities of daily living. Oswestry is scored on a scale of 0-50 with 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
Time Frame: 24 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Foot Orthotic | Sham Orthotic
Number analyzed (Participants) | 21 | 30
units on a scale | 40.3 (13.2) | 37.1 (12.2)

3. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Physical Function
Description: For PROMIS measures, higher scores equals more of the concept being measured (more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. Specifically for PROMIS Physical function 50 indicates the reference population, therefore a score of 40 would be lower physical function.
Time Frame: 24 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Foot Orthotic | Sham Orthotic
Number analyzed (Participants) | 21 | 30
units on a scale | 38.3 (3.9) | 40.9 (4.1)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definitions are consistent with the clinicaltrials.gov definition for adverse, serious adverse event and all cause mortality. In this case there were no deaths in the study and there were no serious adverse events that were determined to be associated with the interventions, therefore this is why the all cause mortality was 0.
Groups:
- Sham Orthotic: Sham Orthotic
  Sham Orthotic: Leather insert without the custom design pads
Arm/Group | Custom Foot Orthotic | Sham Orthotic
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/30
Other Adverse Events (participants affected / at risk) | 0/21 | 0/30

LIMITATIONS AND CAVEATS:
Due to low power secondary to issues with subject recruitment, the findings of this study were inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No